CLINICAL TRIAL: NCT06568627
Title: A Multicenter, Prospective, Randomized, Double Blind, Placebo Controlled, Adaptive Design Study Performed to Evaluate the Efficacy and the Safety of EscharEx in Debridement of Venous Leg Ulcers (VALUE)
Brief Title: A Double Blind Study Performed to Evaluate the Efficacy and the Safety of EscharEx in Debridement of VLU (VALUE)
Acronym: VALUE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MediWound Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MW2022-06-22
Record Dates: First submitted 2024-08-04; First posted 2024-08-23 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Venous Leg Ulcer (VLU)
Keywords: VLU; EscharEx; Debridement; Wound bed preparation
MeSH Terms: conditions — Varicose Ulcer | interventions — Gels

STUDY DESIGN:
Intervention Model Description: A multicenter, prospective, randomized, double blind, placebo controlled, adaptive design study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EscharEx (EX-03) (Active Comparator): EX-03 is the code name of the third generation of EscharEx investigational medicinal product (IMP) formulation. A sterile lyophilized powder containing a concentrate of proteolytic enzymes enriched in bromelain (anacaulase-bcdb ), the active pharmaceutical ingredient (API), that is blended with excipients.
  EX-03 5% powder, should be diluted with Water for Injection (WFI) prior usage.
  Interventions: Drug: EscharEx (EX-03)
- Placebo (Placebo Comparator): Placebo (Gel Vehicle, hydrogel) contains the same excipients as in EX-03, without the API.
  Placebo powder, should be diluted with Water for Injection (WFI) prior usage.
  Interventions: Drug: Placebo (Gel vehicle)

INTERVENTIONS:
Drug: EscharEx (EX-03) — a sterile lyophilized powder containing a concentrate of proteolytic enzymes enriched in bromelain (anacaulase-bcdb). The powder and sterile water are mixed to form a gel prior to application on the wound area.
  Other Names: EX-03
  Arms: EscharEx (EX-03)
Drug: Placebo (Gel vehicle) — A sterile powder containing excipients only (no proteolytic enzymes). The powder and sterile water are mixed to form a gel prior to application on the wound area
  Other Names: Gel vehicle
  Arms: Placebo

SUMMARY:
The main objective of this study is:

To assess the efficacy and safety of EscharEx (EX-03 5% formulation) compared to placebo control,in debridement and wound bed preparation of Venous Leg Ulcers (VLU).

DETAILED DESCRIPTION:
At least 216 eligible adult patients with VLU (with a surface area between 2 cm2 and 25 cm2, and wound age between 4 weeks and 12 months), will be randomized. The patients will be treated with IMP (either EX-03 5% or placebo) in a double blinded manner.

Total duration of the study is up to 27 weeks:

1. Screening period (2 visits, 7 days apart),
2. Daily Visits Period - Debridement with IMP (up to 8 daily site visits within up to 2 weeks),
3. Weekly Visits Period - wound management (up to 11 visits within up to 10 weeks) + optional wound closure confirmation (up to 2 weeks). Wound will be managed in a standardized manner.
4. Monthly Visits Period - Wound Closure Durability Period of 12 weeks starting after wound closure confirmation (3 visits within 12 weeks). per formed only for wound closed during weekly visits period.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, older than 18 years of age,
2. Patients with a VLU (determined by medical history, physical examination, and a documented ultrasound scan demonstrating venous insufficiency),
3. Wound is present for at least 4 weeks but no longer than 1 year,
4. The necrotic/slough/fibrin non-viable tissue area is at least 50% of the wound area (assessed by clinical evaluation),
5. Target wound surface area is in the range of 2-25 cm2 (assessed by eKare inSightTM),
6. Patient understands the nature of the procedure, is able to adhere to the protocol regimen, and provides a written informed consent prior to any study procedure.

Exclusion Criteria:

1. Wound size decreased by > 20% after 1 week of standard-of-care-only period (screening period),
2. Patients with more than one leg ulcer , on the leg of the target wound, with an area greater than or equal to 2 cm2,
3. Signs of clinical infection of the wound or peri-wound, including purulent discharge, deep-tissue abscess, erysipelas, cellulitis, etc.,
4. Severely damaged skin (e.g. abrasion, erosion, exfoliation) extending >2 cm around the wound's edge,
5. Presence of gangrene, signs of systemic infection, sepsis, or osteomyelitis during screening phase,
6. Clinical suspicion of skin cancer (e.g., basal cell carcinoma (BCC), squamous cell carcinoma (SCC), melanoma, or sarcoma), near the target wound, which was not ruled out by biopsy,
7. Patients with skin disorders unrelated to the wound that are presented adjacent to the wound,
8. Patients suffering from chronic skin disorders (Idiopathic Pruritus, Psoriasis, Panniculitis, Pyoderma gangrenosum, etc.) that might deteriorate as a result of local trauma or debridement,
9. Wound has sinus tracts or tunnels extending under healthy tissue or penetrating into periosteum, fascia or bone,
10. Patients with primary lymphatic edema (Lymphedema),
11. A significant decrease in the arterial blood flow of the extremity ,
12. Known small vessels disease (PVD) of any etiology,
13. Patients with pre-enrolment wounds which are covered by eschar heavily saturated with iodine or by silver sulfadiazine (SSD) pseudoeschar (i.e. pseudoeschar as a result of SSD treatment),
14. History of allergy or atopic disease or a known sensitivity to pineapples, bromelain, papaya or papain, as well as known sensitivity to latex proteins (known as latex-fruit syndrome), bee venom or olive tree pollen,
15. Patients with poor nutritional status: albumin < 2.5g/dl, poorly controlled diabetes Mellitus (HbA1c > 12%), anemia (hemoglobin<8 g/dL), a leukocyte counts < 3,000/μl or >15000/μl, neutrophil count ≤1000/ μl, platelets <100,000/μl, abnormal liver function (AST, ALT>2 x upper limit of normal range), renal failure (Cr > 2.5 mg/dl and eGFR < 30ml/ min /1.73m2), BMI>48,
16. INR>2 or PTT > x 2 ULN (unless the patient receives coumarin derivatives anticoagulants (e.g. warfarin), and the INR and PTT levels are in their required levels and are stable),
17. Patients undergoing renal or peritoneal dialysis,
18. Any condition that would preclude safe participation in the study, e.g. significant or unstable cardiovascular, pulmonary, liver, hematological, immunological, neoplastic disease, active COVID-19, or any immediate life threatening condition,
19. Recent history or concurrent acute injury or disease that might compromise the patient's welfare, according to investigator discretion,
20. Patient is currently receiving, or has received at any time within three months prior to enrollment, or is planned to receive during trial period, any medications or treatments known to affect the wound healing processes; these include chronic systemic steroid intake with topical skin changes (i.e. thin, fragile skin with multiple heamatomas or previous laceration history) immuno-suppressive drugs, immunomodulating medications, chemotherapy and radiation therapy,
21. In case the subject is treated with Pentoxifylline, dosing is stable less than 4 weeks,
22. Mentally incompetent adults who are incapable of giving legal consent (e.g. dementia, psychiatric patients, etc.),
23. Concurrent use of non-approved drugs or alcohol abuse,
24. Pregnant women (positive pregnancy test) or nursing mothers,
25. Exposure to investigational intervention within three months prior to enrollment, or anticipated participation in another investigational drug trial or other intervention trial, while enrolled in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of complete debridement, clinically (visually) assessed after each application | up to 2 weeks
  counting events of complete debridement
Incidence of complete wound closure | up to 12 weeks
  counting events of complete wound closure

SECONDARY OUTCOMES:
Incidence of complete healthy viable granulation tissue, as assessed clinically | up to 2 weeks
  counting events of complete granulation
Time to the first declaration of complete debridement, clinically assessed | up to 12 weeks
  count in days
Time to complete wound closure, clinically assessed | up to 12 weeks
  count in days
Percent change in wound area, as assessed by eKare inSightTM | up to 12 weeks
  count in percentage

OTHER OUTCOMES:
Incidence and severity of systemic and local adverse events | up to 27 weeks
Incidence of target wound infections | up to 27 weeks
  counting events
Incidence of discontinuation due to adverse events | up to 27 weeks
  counting events of discontinuation
Change in pain, as assessed by Numeric Pain Rating Scale (NPRS) | up to 12 weeks
Immunogenicity evaluation | baseline, post last daily visit, 4 and 10 weeks following last daily visit, and on last monthly visit
  measurement of Anti-Drug-Antibodies levels

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Limb Preservation Platform, Inc, Fresno, California
  - Center for Clinical Research INC, San Francisco, California
  - Northwell Health Comprehensive Wound Healing Center, Lake Success, New York
  - JPS Health Network/Acclaim Multispecialty Clinic, Fort Worth, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No